CLINICAL TRIAL: NCT03826199
Title: Evaluation of Pre-exposure Prophylaxis Cascade in Pregnant and Breastfeeding Women in Cape Town, South Africa (Formative Study)
Brief Title: Evaluation of Pre-exposure Prophylaxis Cascade in Pregnant and Breastfeeding Women in Cape Town (Formative Study)
Acronym: PrEP-PP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of Cape Town (Other); Desmond Tutu HIV Foundation (Other)
Responsible Party: Principal Investigator, Dvora Joseph Davey, PhD, MPH, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: K01TW011187 (NIH)
Record Dates: First submitted 2019-01-25; First posted 2019-02-01 (Actual); Results first posted 2023-03-16 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Hiv
Keywords: pre-exposure prophylaxis; PrEP; pregnancy; prevention of mother to child transmission; PMTCT
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Prenatal Care; Postnatal Care

STUDY DESIGN:
Intervention Model Description: Open label cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: TDF-FTC — We will investigate the feasibility and acceptability of integrating PrEP into antenatal and postnatal/well-baby services. Upon enrollment in the cascade, all women will be offered PrEP counseling and information, and patients will be followed regardless of their choice to initiate PrEP or not. Participants who initiate PrEP will receive TDF-FTC during the study. At each study visit (every 3-months), women will receive counseling on PrEP adherence or on the risks and benefits of PrEP for women not yet initiated. We will evaluate PrEP initiation and adherence in pregnant and breastfeeding women (N=220) from first antenatal care visit through 12 months post-partum.
  Other Names: PrEP; Truvada
Behavioral: Counselling on PrEP in antenatal and postnatal care — Information about PrEP will be integrated into regular group education in ANC by existing health care providers during discussion about HIV testing and treatment. During every study visit, PrEP counseling (including adherence counseling for women already on PrEP) will be provided. For women not on PrEP, counselling will be provided on PrEP and HIV prevention.

SUMMARY:
The overarching goal of this proposal is to evaluate the feasibility and acceptability of integrating PrEP into antenatal and postnatal care, to describe the cascade in women initiating PrEP in this setting, and to evaluate the reasons for attrition along the PrEP cascade in a cohort of pregnant and breastfeeding women. The specific aims are to: (1) Evaluate the feasibility and acceptability of integrating PrEP into antenatal and postnatal/well-baby services; (2) Describe the PrEP cascade of initiation, retention, and adherence in a cohort of 220 HIV-uninfected pregnant and breastfeeding women, (3) Evaluate attrition and associated factors across the PrEP cascade.

ELIGIBILITY:
Inclusion Criteria:

1. Documented HIV-negative according to two fingerpick rapid tests (per routine antenatal care protocol in this setting), confirmed with a 4th generation antigen HIV test at study enrollment
2. No previous exposure triple-drug antiretroviral therapy
3. Age 18 years or older
4. Lives within 20 kilometers of a clinic
5. Without psychiatric or medical contraindications to PrEP use
6. Able to provide informed consent for research

Exclusion Criteria:

Failure to meet any of the inclusion criteria

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Only pregnant women will be included
Enrollment: 200 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Gugulethu Midwife Obstetric Unit, Cape Town, South Africa

REFERENCES:
- [Background] Joseph Davey D, Myer L, Coates T. PrEP implementation in pregnant and post-partum women. Lancet HIV. 2020 Jan;7(1):e5-e6. doi: 10.1016/S2352-3018(19)30371-6. Epub 2019 Dec 5. No abstract available. PMID 31813838
- [Result] Khadka N, Gorbach PM, Nyemba DC, Mvududu R, Mashele N, Javanbakht M, Nianogo RA, Aldrovandi GM, Bekker LG, Coates TJ, Myer L, Joseph Davey DL. Evaluating the use of oral pre-exposure prophylaxis among pregnant and postpartum adolescent girls and young women in Cape Town, South Africa. Front Reprod Health. 2023 Sep 19;5:1224474. doi: 10.3389/frph.2023.1224474. eCollection 2023. PMID 37795521
- [Result] Joseph Davey DL, Knight L, Markt-Maloney J, Tsawe N, Gomba Y, Mashele N, Dovel K, Gorbach P, Bekker LG, Coates TJ, Myer L. "I had Made the Decision, and No One was Going to Stop Me" -Facilitators of PrEP Adherence During Pregnancy and Postpartum in Cape Town, South Africa. AIDS Behav. 2021 Dec;25(12):3978-3986. doi: 10.1007/s10461-021-03320-x. Epub 2021 Jun 3. PMID 34085132
- [Result] Joseph Davey DL, Mvududu R, Mashele N, Lesosky M, Khadka N, Bekker LG, Gorbach P, Coates TJ, Myer L. Early pre-exposure prophylaxis (PrEP) initiation and continuation among pregnant and postpartum women in antenatal care in Cape Town, South Africa. J Int AIDS Soc. 2022 Feb;25(2):e25866. doi: 10.1002/jia2.25866. PMID 35138678
- [Result] Moran A, Mashele N, Mvududu R, Gorbach P, Bekker LG, Coates TJ, Myer L, Joseph Davey D. Maternal PrEP Use in HIV-Uninfected Pregnant Women in South Africa: Role of Stigma in PrEP Initiation, Retention and Adherence. AIDS Behav. 2022 Jan;26(1):205-217. doi: 10.1007/s10461-021-03374-x. Epub 2021 Jul 21. PMID 34287756
- [Result] Haribhai S, Khadka N, Mvududu R, Mashele N, Bekker LG, Gorbach P, Coates TJ, Myer L, Joseph Davey DL. Psychosocial determinants of pre-exposure prophylaxis use among pregnant adolescent girls and young women in Cape Town, South Africa: A qualitative study. Int J STD AIDS. 2023 Jul;34(8):548-556. doi: 10.1177/09564624231152776. Epub 2023 Mar 22. PMID 36947792

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregnant Women Offered PrEP: Pregnant women in antenatal care (16+ years) were offered oral TDF/FTC as PrEP in a cohort study
Period: Overall Study
Arm/Group | Pregnant Women Offered PrEP
Started | 200
Completed | 200
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 200 pregnant women enrolled in formative study and followed for 12 months postpartum
Arm/Group | Pregnant Women Offered PrEP
Number analyzed (Participants) | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 190
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 25 [22 to 32]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 200
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 200
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 200

OUTCOME MEASURES:

1. Primary Outcome: PrEP Retention
Description: number of women on PrEP who return for study visits (do not miss more than 1 visit) / total number of women in active cohort who are prescribed PrEP
Time Frame: 18 months
Population: Participants who were retained on PrEP study and were on PrEP
Measure: Number; unit: participants
Arm/Group | Pregnant Women Offered PrEP
Number analyzed (Participants) | 200
participants | 100

2. Primary Outcome: PrEP Adherence
Description: number of women taking PrEP who have >80 percent levels at >40ng/mL tenofovir diphosphate (indicating dosing in past 24 hours) / total woman-time on PrEP in active cohort = PrEP adherence rate (objective)
Time Frame: 3 months
Population: Women who were adherent on PrEP at 3 months per DBS measure of TFV-DP (equivalent to 2+ days/week by pregnant or postpartum)
Measure: Number; unit: participants
Arm/Group | Pregnant Women Offered PrEP
Number analyzed (Participants) | 78
participants | 25

3. Secondary Outcome: PrEP Initiation
Description: number of women who initiate PrEP over time/ total number of women in active cohort
Time Frame: 18 months
Population: Pregnant women who enrolled in study and were offered PrEP
Measure: Count of Participants; unit: Participants
Arm/Group | Pregnant Women Offered PrEP
Number analyzed (Participants) | 200
Participants | 180

4. Secondary Outcome: PrEP Adherence (Peri-sexual)
Description: number of women taking PrEP who have >80 percent levels at >40ng/mL tenofovir diphosphate (indicating dosing in past 24 hours) / total woman-time when women report condomless sex in past week= PrEP adherence rate (peri-sexual)
Time Frame: 3 months
Population: 78 DBS drawn from participants on PrEP at 3m visit
Measure: Count of Participants; unit: Participants
Arm/Group | Pregnant Women Offered PrEP
Number analyzed (Participants) | 78
Participants | 25

5. Secondary Outcome: PrEP Adherence (Subjective, Self-reported)
Description: number of women taking PrEP, who self-report taking their medication daily (and pill count to confirm this) during periods of sexual risk over time / total woman time on PrEP in active cohort = PrEP adherence rate (subjective)
Time Frame: 3 months
Population: Participants who started PrEP at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Pregnant Women Offered PrEP
Number analyzed (Participants) | 194
Participants | 118

ADVERSE EVENTS:
Time Frame: We collected data every study visit (quarterly) until 12 months postpartum (up to 18 months from baseline enrollment in study)
Description: Adverse events included all pregnancy and birth outcomes in the cohort
Arm/Group | Pregnant Women Offered PrEP
All-Cause Mortality (participants affected / at risk) | 0/200
Serious Adverse Events (participants affected / at risk) | 10/200
Other Adverse Events (participants affected / at risk) | 0/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregnant Women Offered PrEP (N=200)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 1 (1) — Pregnancy loss at >20 weeks gestation
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 5 (5) — Pregnancy loss at <=20 weeks gestation
Infant low birthweight or preterm (Pregnancy, puerperium and perinatal conditions) | 4 (4) — LBW <2500 grams; preterm born <37 weeks gestation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-11): https://cdn.clinicaltrials.gov/large-docs/99/NCT03826199/Prot_SAP_000.pdf